CLINICAL TRIAL: NCT00134290
Title: The Effects of Calorie Restriction - Whether or Not Calculated Based on BMR (Basic Metabolic Rate) - With or Without Metformin on Weight and Insulin Resistance of Obese Insulin Resistant Patients
Brief Title: The Effects of Calorie Restriction With or Without Metformin on Weight and Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002/032
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Body Weight; Insulin Resistance
MeSH Terms: conditions — Body Weight; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: metformin
Behavioral: "standard diet advice"
Behavioral: "personal diet advice"

SUMMARY:
This is a study to:

* Determine the difference between strong hypo-energetic "standard diet advice" and modest hypo-energetic "personal diet advice"; and
* Determine the influence of insulin-insensitivity on obesity and weight reduction by treating patients with metformin or placebo.

DETAILED DESCRIPTION:
The aim of the present study was to determine what the difference is of a strong hypo-energetic "standard diet advice" and a modest hypo-energetic "personal diet advice" which was determined by the energy needs of a person as calculated with a combination of basal metabolic rate (BMR) and physical activity level (PAL) on weight loss and insulin sensitivity.

Secondly, this study wanted to determine what the influence is of insulin-insensitivity on obesity and weight reduction by treating the patients with metformin or placebo. The subjects were therefore randomised into two double blinded groups receiving either metformin (2 x 850 mg per day) or placebo in combination with a moderate energy restriction and a exercise regimen of 30 minutes per day for 1 year.

Treatment effects of both diets and the effect of metformin on weight reduction and insulin sensitivity were determined after a treatment period of 20 and 52 weeks.

Insulin sensitivity was quantified using the homeostasis model assessment (HOMA) and the OGTT. Body composition was determined with the bioelectrical impedance method.

Blood was also drawn for hormonal and biochemical analyses after 20 and 52 weeks of treatment. Furthermore, the patients had to fill out a 3-day food diary at baseline, after 20 weeks and after 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 20-55 years of age
* Body mass index (BMI) equal to or greater than 30 kg/m²
* Insulin resistance as determined by oral glucose tolerance test (OGTT) and HOMA

Exclusion Criteria:

* Diabetes mellitus, kidney insufficiency, or hepatic insufficiency
* Hypogonadism with other etiology than overweight
* Pregnancy
* BMI equal to or greater than 40 kg/m²

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48
Dates: Start 2002-01; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Effect of diet on weight and insulin sensitivity/insulin resistance after 20 and 52 weeks of treatment

SECONDARY OUTCOMES:
Effect of metformin on weight and insulin resistance after 20 and 52 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Giri, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be